CLINICAL TRIAL: NCT01939665
Title: PANFIRE - Pilot-study: Non-thermal Ablation Using Irreversible Electroporation (IRE) to Treat Locally Advanced Pancreatic Carcinoma - a Phase I Clinical Trial
Brief Title: PANFIRE Study: Irreversible Electroporation (IRE) to Treat Locally Advanced Pancreatic Carcinoma
Acronym: PANFIRE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. M.R. Meijerink, Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL42888.029.13; 2013/155 (Registry Identifier: 2013/155)
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced Pancreatic Carcinoma (LAPC); Non-metastasized Unresectable Pancreatic Carcinoma; Pancreatic Cancer
Keywords: Locally advanced pancreatic carcinoma; LAPC; Irreversible electroporation; NanoKnife; IRE; Safety; Efficacy; Non-thermal ablation; Percutaneous ablation; Low Energy Direct Current
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irreversible electroporation (Experimental): Single arm study: Percutaneous irreversible electroporation of locally advanced pancreatic carcinoma
  Interventions: Device: NanoKnife "Irreversible electroporation (IRE)"

INTERVENTIONS:
Device: NanoKnife "Irreversible electroporation (IRE)" — Tumor ablation with irreversible electroporation with the NanoKnife
  Other Names: IRE; NanoKnife

SUMMARY:
Irreversible electroporation (IRE) is a new, minimal-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels and bile ducts. With IRE, multiple electrical pulses are applied to tumorous tissue. These pulses alter the existing transmembrane potential of the cell membranes, and create 'nanopores', after which the cell dies through loss of homeostasis.

The purpose of this study is to investigate the safety of percutaneous IRE in the treatment of patients with locally advanced pancreatic carcinoma (LAPC). Other objectives are feasibility and efficacy of IRE based upon symptomatic response and tumor response.

Fourty patients with histologically confirmed locally advanced pancreatic adenocarcinoma (<5cm) will undergo percutaneous irreversible electroporation of the tumor using CT and ultrasound guidance. After IRE, patients will be carefully monitored and any (serious) adverse events are registered. Follow-up will consist of frequent CT scanning, as well as serum CA19.9 tumor marker.

We hypothesize that IRE in the pancreas will induce good symptom palliation and local tumor control, without causing severe complications.

ELIGIBILITY:
Inclusion Criteria:

Screening must be performed no longer than 2 weeks prior to study inclusion.

* Radiologic confirmation of LAPC by at least ceCT of chest and abdomen (with the upper abdomen scanned according to a dedicated 3mm slice multiphase pancreatic tumor protocol), performed maximum 2 weeks prior to the procedure;
* Maximum tumor diameter ≤ 5 cm;
* Histological or cytological confirmation of pancreatic adenocarcinoma;
* Age ≥ 18 years;
* ASA-classification 0 - 3
* Life expectancy of at least 12 weeks;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to definite inclusion;

  * Hemoglobin ≥ 5.6 mmol/L;
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3;
  * Platelet count ≥ 100*109/l;
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * ALT and AST ≤ 2.5 x ULN;
  * Serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 50 ml/min;
  * Prothrombin time or INR < 1.5 x ULN;
  * Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed if this treatment can be interrupted as judged by the treating physician);
* Written informed consent;

Exclusion Criteria:

* Resectable pancreatic adenocarcinoma as discussed by our multidisciplinary hepatobiliary team;
* Extrapancreatic metastases;
* Successful down staging after (radio)chemotherapy from previous unresectable/borderline tumor to resectable tumor;
* Stage IV pancreatic carcinoma;
* History of epilepsy;
* History of cardiac disease:

  * Congestive heart failure >NYHA class 2;
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening);
  * Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers for antihypertensive regimen are permitted);
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0);
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment;
* Immunotherapy ≤ 6 weeks prior to the procedure;
* Chemotherapy ≤ 6 weeks prior to the procedure;
* Radiotherapy ≤ 6 weeks prior to the procedure;
* Concomitant use of anti-convulsive and anti-arrhythmic drugs (other than beta blockers used for antihypertensive);
* Allergy to contrast media;
* Any implanted stimulation device;
* Any implanted metal stent/device within the area of ablation that cannot be removed;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study;

Of note, patients with contra-indications for MRI will not be excluded from participation: in this case radiologic follow-up will consist of CT-scanning according to protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Safety (number of adverse events) | early: 90 days; late: 12 months
  Number of adverse events of IRE-treatment (within 12 months after treatment) are registered and analyzed according to the CTCAE version 4.0. Complications related to IRE are early complications during hospital admission (e.g. bile leak, bowel leak, infection, pancreatitis), or late complications of IRE such as bile duct stenosis that become apparent during follow-up in the year after treatment.

SECONDARY OUTCOMES:
Tumor response | 12 months
  * Ablation success: the ability to deliver the planned therapy and at 3 months to have no evidence of residual tumor;
  * Local recurrence rate (LRR): defined as the reappearance of viable tumor after a period of time during which viable tumor could not be detected;
  * Overall survival and (local and distant) progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R Meijerink, MD, PhD, Principal Investigator — VU University Medical Center, Department of Radiology and Nuclear Medicine; Geert Kazemier, Prof. Dr., Principal Investigator — VU University Medical Center, Department of Surgery; Cornelis van Kuijk, Prof. Dr., Study Director — VU University Medical Center, Head of Department of Radiology,
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Ruarus AH, Vroomen LGPH, Geboers B, van Veldhuisen E, Puijk RS, Nieuwenhuizen S, Besselink MG, Zonderhuis BM, Kazemier G, de Gruijl TD, van Lienden KP, de Vries JJJ, Scheffer HJ, Meijerink MR. Percutaneous Irreversible Electroporation in Locally Advanced and Recurrent Pancreatic Cancer (PANFIRE-2): A Multicenter, Prospective, Single-Arm, Phase II Study. Radiology. 2020 Jan;294(1):212-220. doi: 10.1148/radiol.2019191109. Epub 2019 Nov 5. PMID 31687922
- [Derived] Witvliet-van Nierop JE, Lochtenberg-Potjes CM, Wierdsma NJ, Scheffer HJ, Kazemier G, Ottens-Oussoren K, Meijerink MR, de van der Schueren MAE. Assessment of Nutritional Status, Digestion and Absorption, and Quality of Life in Patients with Locally Advanced Pancreatic Cancer. Gastroenterol Res Pract. 2017;2017:6193765. doi: 10.1155/2017/6193765. Epub 2017 Aug 20. PMID 28912804